CLINICAL TRIAL: NCT00083980
Title: KAVA KAVA in Generalized Anxiety: A Double-Blind Trial
Brief Title: Kava Kava for the Treatment of Generalized Anxiety Disorder (GAD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: European reports of liver toxicity from kava meant that the study had to stop
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01AT000150-01A1 (NIH)
Record Dates: First submitted 2004-06-04; First posted 2004-06-07 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2006-08

CONDITIONS: Anxiety Disorders
Keywords: Kava; Complementary Therapies; Medicine, Herbal
MeSH Terms: conditions — Anxiety Disorders | interventions — Venlafaxine Hydrochloride; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- active antidepressant drug comparator (Active Comparator): Venlafaxine ER
  Interventions: Drug: Venlafaxine ER; Drug: Sugar pill
- Sugar pill (Placebo Comparator): Inert placebo pills as duble dummy - up to 4 per day for kava and 3 per day for venlafaxine
  Interventions: Drug: Sugar pill
- Herbal treatment kava (Experimental): Kava
  Interventions: Drug: Sugar pill; Drug: Kava

INTERVENTIONS:
Drug: Venlafaxine ER — 75 to 225 mg daily
  Other Names: Effexor XR
  Arms: active antidepressant drug comparator
Drug: Sugar pill — Upto 3 per day for venlafainxe and 4 per day for kava placebos.
  Other Names: No brand name
Drug: Kava — 140 to 280 mg per day
  Other Names: No brand name
  Arms: Herbal treatment kava

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the herbal medicine kava kava for the treatment of generalized anxiety disorder (GAD).

DETAILED DESCRIPTION:
Kava kava (KAV) is a plant-derived treatment widely used in Europe to treat anxiety disorders. Several studies suggest that KAV may be effective in reducing anxiety symptoms; however, trial data are limited. This study will compare KAV, the drug venlafaxine-XR (VEN), and placebo for the treatment of GAD.

This study will last 10 weeks. Participants will be randomly assigned to receive KAV, VEN, or placebo for 8 weeks. Participants will then undergo a 1-week tapering of their medication followed by an additional week of observation. Self-report scales and questionnaires will be used to assess the anxiety, depression, and functional impairment of participants. Side effects, vital signs, and laboratory measures will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of generalized anxiety disorder (GAD)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2002-06; Primary Completion 2004-06 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Hamilton Anxiety Scale | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Davidson, MD, Principal Investigator — Duke University